CLINICAL TRIAL: NCT00418899
Title: Gliogene: Brain Tumor Linkage Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2003-0974; 1R01CA119215-01A1 (NIH)
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Brain Tumor; Glioma
Keywords: Brain Tumor; Glioma; Linkage Study; Survey; Gliogene; High-risk familial brain tumor pedigrees
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — About 3 tablespoons of blood will be drawn and if unable to donate blood, researchers will collect a saliva sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLIOGENE: International Multi-Center, Multidisciplinary Study Consortium
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire, 30-40 minutes, about gliomas and its risk factors (such as environmental and genetic information).
  Other Names: Survey

SUMMARY:
The goal of this research study is to investigate the role of genes that may point to a higher risk of developing a glioma. Researchers will use new gene mapping techniques to study how high-risk factors are passed on through a family's genes and increase the risk of developing gliomas.

Objectives:

We propose an international multi-center, multidisciplinary study consortium, GLIOGENE, to identify susceptibility genes in high-risk familial brain tumor pedigrees using the most sophisticated genetic analysis methods available. To address our hypothesis, we propose the following specific aims:

Aim 1: Establish a cohort of 400 high-risk pedigrees for genetic linkage analysis. To date, we have identified and collected biologic samples from 20 high-risk families that have met our criteria of 2 or more relatives diagnosed with a brain tumor. From the 15 centers in the United States and Europe, we will screen and obtain epidemiologic data from approximately 17,080 gliomas cases to identify a target of 400 families for genetic analysis. We will establish a cohort of the first and second-degree relatives from these glioma cases to obtain new knowledge about how cancer aggregates in glioma families. We will also acquire biospecimens (blood and tumor tissue), and risk factor data from relevant family members.

Aim 2: Identify candidate regions linked to familial brain tumors. To strengthen evidence of linkage to regions found in our preliminary analysis and to identify additional regions linked to brain tumors, we will genotype informative glioma pedigrees identified in aim 1 using Affymetrix 10K GeneChip with markers spaced throughout the genome, and conduct a genome-wide multipoint linkage scan with these markers.

Aim 3: Fine map the regions established in Aim 2 by genotyping selected SNPs from genome databases. We will attempt to further refine the regions identified in Aim 2 to less than 1cM by using approximately 1,500 - 2,000 carefully selected SNPs. The prioritization of regions will be based on a combination of the strength of evidence for linkage from families of various ethnic backgrounds and the presence of obvious candidate genes.

DETAILED DESCRIPTION:
A consortium (group) of researchers wants to learn more about gliomas as well as the risk factors (such as environmental and genetic information) for patients with this kind of brain tumor. Participants in this study will be part of a glioma genetic epidemiology study (herein referred to as "GLIOGENE") involving eleven centers in the United States (U.S.) and five centers in Europe. The eleven centers in the U.S. are: The University of Texas MD Anderson Cancer Center (MD Anderson); Baylor College of Medicine, Texas Children's Hospital (TCH); Brigham and Women's Hospital (BWH); Case Western Reserve University (CWRU); Columbia University Medical Center (CUMD); Duke University (Duke); Mayo Clinic Rochester (Mayo); Memorial Sloan-Kettering Cancer Center (MSKCC); University of California, San Francisco (UCSF); University of Illinois, Chicago (UIC); and Evanston Northwest Healthcare (ENWH). The five centers in Europe are: Gertner Institute, Israel (Gertner); Institute of Cancer Epidemiology, Denmark (ICE); Institute of Cancer Research (ICR), United Kingdom (U.K.); Tampere University Hospital (TU) and Umeå University Hospital, Sweden (Umeå).

If you agree to take part in this study, you will have about 3 tablespoons of blood drawn. If you are unable to donate blood, researchers will collect a saliva sample.

In addition, if you have 2 or more family members with a glioma, a trained research interviewer will ask you questions using a questionnaire that will take about 30-40 minutes to complete. The topics in the questionnaire will include demographic data (such as age and race), environmental exposures, medical history, family history of cancer and other conditions, and other lifestyle factors.

Study staff will only use any names and contact information of relatives or other potential research participants provided to MD Anderson in order to contact those individuals to find out if they are eligible and desire to participate in this study.

Before your blood and/or saliva is sent to TCH for banking, your name and any personal identifying information will be coded to protect your privacy. MD Anderson will not have oversight of any leftover blood and/or saliva that will be banked by THC for additional research. Blood and saliva that are collected will only be used by researchers involved in this study.

Neither you nor your physicians will receive individual reports of this research. Results will not be placed in your health records. All information will be kept confidential and used only for research purposes. For the results, your sample, contact and medical information will be linked by assigning an identification number (instead of your name).

In the event that any participant has participated in prior glioma studies conducted by Melissa L. Bondy (ID00-098 or ID 91-036), signing the informed consent for this study will allow us to use their specimens previously collected.

There is a rare chance that a research team member could be accidentally exposed to your blood or body fluids. If that occurs, extra blood (about 2 teaspoons) may be drawn to test for infections such as hepatitis and HIV (the AIDS virus). An existing blood sample may be used for these tests instead. You will be told that your blood is being tested and the results of your test. Researchers will ask how you would like to receive the results, such as by phone or certified letter. The test results and your name, address, date of birth, and sex will be recorded in the confidential MD Anderson medical records.

If you test positive for hepatitis or HIV, the test results and your name, address, date of birth, and sex will be shared with appropriate health authorities as required by law. You will also be given a list of places in your area so that you can receive further testing and treatment.

Your participation will be over in this study after the data has been collected and finalized.

This is an investigational study. Up to 17,080 participants will take part in this multicenter study. Up to 9,000 will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) An affected or unaffected member of a family that has two or more reported gliomas (ICD9 codes 191.0-191.9) in the family.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with a glioma or a family member of someone with a glioma.
Sampling Method: Non-Probability Sample
Enrollment: 17080 (Estimated)
Dates: Start 2004-02-12 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Patients' Susceptibility Genes in High-risk Familial Brain Tumor Pedigrees | 13 Years (Collection of blood tests and survey/interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Shete, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (15):
- United States (10):
  - University of California Medical Center, San Francisco, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Medical Center, Chicago, Chicago, Illinois
  - Evanston NW Healthcare, Evanston, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Institute of Cancer Epidemiology, Copenhagen, Denmark
- Tampere University Hospital, Tampere, Finland
- The Danek Gertner Institute, Tel Litwinsky, Israel
- Umeå University Hospital, Umeå, Sweden
- Institute of Cancer Research, London, United Kingdom

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org